CLINICAL TRIAL: NCT07277972
Title: An Open-Label, Single-Arm, Multicenter, Phase II Clinical Study of Iparomlimab and Tuvonralimab Injection in Combination With Lenvatinib or Axitinib for the Treatment of Locally Advanced or Metastatic Clear Cell Renal Cell Carcinoma That Has Failed First-Line Systemic Therapy
Brief Title: Iparomlimab and Tuvonralimab Injection in Combination With Lenvatinib or Axitinib for the Treatment of Locally Advanced or Metastatic Clear Cell Renal Cell Carcinoma That Has Failed First-Line Systemic Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20251137
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: RCC, Renal Cell Cancer
Keywords: lparomlimab and Tuvonralimab Injection; Lenvatinib; Axitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab Injection in combination with Lenvatinib or Axitinib (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection in combination with Lenvatinib or Axitinib

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection in combination with Lenvatinib or Axitinib — Iparomlimab and Tuvonralimab Injection: 5 mg/kg, iv, q3w, for a cumulative maximum treatment duration of 2 years; Lenvatinib: Starting dose of 12 mg, po, qd, q3w; or Axitinib: 5 mg, po, bid, q3w.

SUMMARY:
The primary objective is to evaluate the improvement in Objective Response Rate (ORR) achieved with Iparomlimab and Tuvonralimab Injection (QL1706, an Anti-PD-1/CTLA-4 Combined Antibody) in combination with Lenvatinib or Axitinib, in patients with locally advanced or metastatic clear cell renal cell carcinoma (ccRCC) who have failed first-line systemic therapy.

DETAILED DESCRIPTION:
This single-arm, multicenter clinical study aims to evaluate the improvement in Objective Response Rate (ORR) achieved with Iparomlimab and Tuvonralimab Injection (QL1706, an Anti-PD-1/CTLA-4 Combined Antibody) in combination with Lenvatinib or Axitinib, in patients with locally advanced or metastatic clear cell renal cell carcinoma (ccRCC) who have failed first-line systemic therapy.This study consists of three phases: screening, treatment, and follow-up.Efficacy evaluation and safety monitoring should be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age at Diagnosis: ≥18 years.
* Histologically confirmed locally advanced or metastatic clear cell renal cell carcinoma.
* Disease progression or intolerance during or following first-line systemic therapy.
* ECOG Performance Status: 0-1.
* At least one measurable lesion as defined by RECIST v1.1.
* Life expectancy ≥12 weeks.
* Adequate bone marrow function: White blood cell count > 4.0×10⁹/L, Hemoglobin > 90 g/L, Platelet count > 100×10⁹/L.
* Adequate hepatic and renal function: Total bilirubin ≤ 1.5 × ULN; Aspartate aminotransferase and/or Alanine aminotransferase ≤ 2.5 × ULN; Alkaline phosphatase ≤ 2.5 × ULN; Serum creatinine ≤ 1.5 × ULN.
* Adequate coagulation function: International Normalized Ratio (INR) ≤1.5 × ULN, Activated Partial Thromboplastin Time (APTT) ≤1.5 × ULN.
* The patient must provide signed informed consent and be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures as specified in the study protocol.
* Female subjects of childbearing potential must agree to use reliable contraceptive methods (e.g., condoms, prescribed oral contraceptives taken regularly) from screening until 1 year after the end of treatment.

Exclusion Criteria:

* Allergy to any component of macromolecular protein preparations; contraindications or hypersensitivity to any ingredient of Iparomlimab and Tuvonralimab Injection, Lenvatinib, or Axitinib.
* Major surgery within 28 days prior to the first dose (excluding diagnostic laparoscopy; local surgery for isolated lesions is acceptable).
* Positive Hepatitis B surface antigen (HBsAg) with HBV DNA >1×10³ copies/mL, or positive anti-Hepatitis C virus (HCV) antibody.
* Positive anti-HIV antibody or a diagnosis of Acquired Immunodeficiency Syndrome (AIDS).
* Active, known, or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary disorders, nephritis, vasculitis, systemic lupus erythematosus, hyperthyroidism, hypothyroidism, asthma requiring bronchodilator therapy). Exceptions include type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy only, and skin disorders not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
* Renal failure requiring hemodialysis or peritoneal dialysis.
* History of interstitial lung disease (ILD) or pneumonitis requiring oral or intravenous steroids within the past year; administration of Vancomycin within the past month.
* Chronic systemic glucocorticoid therapy (at a dose equivalent to ≥10 mg prednisone daily) or any other form of immunosuppressive therapy. Subjects using inhaled or topical corticosteroids are eligible.
* Uncontrolled cardiac disease, such as: 1) Heart failure, NYHA class ≥ II; 2) Unstable angina; 3) Myocardial infarction within the past year; 4) Supraventricular or ventricular arrhythmia requiring treatment or intervention.
* Thromboembolic events within 6 months prior to the start of study treatment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), or pulmonary embolism, etc.
* Known central nervous system metastases.
* Urinalysis indicating urine protein ≥ +++ and confirmed 24-hour urinary protein >1.0 g.
* Pregnant or lactating women (a pregnancy test should be considered for sexually active women of childbearing potential).
* Prior or concurrent other malignancies, except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary carcinoma of the thyroid.
* Active infection requiring systemic therapy within one week.
* Administration of a live vaccine within 30 days prior to the first dose of Iparomlimab and Tuvonralimab Injection.
* History of organ transplantation or hematopoietic stem cell transplantation.
* Any other condition that, in the investigator's assessment, may compromise patient safety or compliance, such as severe concomitant illnesses (including psychiatric disorders) requiring prompt treatment, severely abnormal laboratory test results, or the presence of other psychological, familial, or sociogeographic factors posing high-risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 12 month
  the percentage of participants in the analysis population who had a CR(Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 12 month
  PFS was defined as the time from first dose of study treatment to the first documented PD per REClST 1.1 by investigator assessment, or death due to any cause, whichever occurred first.
Duration of Response | up to 12 month
  For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigator assessment, DOR was defined as time from first documented CR or PR until PD or death，whichever occurs first.
Overall survival | up to 36 month
  OS was defined as the time from the first dose of study drug to death due to any cause.
Adverse Events | up to 36 month
  An AE was defined as any untoward medical occurrence in a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yao, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

IPD SHARING:
Plan to Share IPD: No